CLINICAL TRIAL: NCT00273858
Title: Open Label Study To Evaluate The Safety Profile And The Quality Of Life In Patients Receiving Etanercept For The Treatment Of Rheumatoid Arthritis, Ankylosing Spondylitis And Psoriatic Arthritis
Brief Title: Study Evaluating the Safety of Etanercept in Rheumatoid Arthritis, Ankylosing Spondylitis and Psoriatic Arthritis
Status: Terminated | Type: Observational
Why Stopped: The study was terminated because at least one year follow-up was achieved for each patient and the achievement of 965 exposure years to the drug.
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881A-101695; B1801106
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Results first posted 2011-07-28 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: Ankylosing Spondylitis; Arthritis, Psoriatic; Arthritis, Rheumatoid; Spondylitis, Ankylosing
Keywords: Rheumatoid Arthritis; Ankylosing Spondylitis; Psoriatic Arthritis
MeSH Terms: conditions — Spondylitis, Ankylosing; Arthritis, Psoriatic; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- etanercept: Patients already prescribed to receive etanercept for the first time for treatment of Rheumatoid Arthritis, Ankylosing Spondylitis or Psoriatic Arthritis according to the Summary of Product Characteristics (SmPC).
  Interventions: Other: There is no Intervention. The study is observational.

INTERVENTIONS:
Other: There is no Intervention. The study is observational. — The study is observational and the prescription follows the SmPC of etanercept.

SUMMARY:
This is a Phase 4 open label, non-interventional, multi-center study to evaluate the safety of Enbrel (etanercept) treatment in patients receiving etanercept 25mg sc twice weekly or 50mg of etanercept once weekly. The improvement of health-related quality of life will also be evaluated.

DETAILED DESCRIPTION:
Patients already prescribed to receive etanercept for the first time for treatment of Rheumatoid Arthritis, Ankylosing Spondylitis or Psoriatic Arthritis according to the Summary of Product Characteristics (SmPC).

Patients have been recruited sequentially based on eligibility criteria up to the number limit assigned to each site.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at time of consent
* Satisfies the 1987 ACR Revised Criteria for Rheumatoid Arthritis or has a diagnosis of ankylosing spondylitis or psoriatic arthritis, as determined by the doctor
* Provides informed consent
* Demonstrate a negative serum or urine pregnancy test prior to administration of etanercept. Sexually active women participating in the study must use a medically acceptable form of contraception.
* Patients already prescribed etanercept according to approved labelling

Exclusion Criteria:

* Has hypersensitivity to etanercept
* Has sepsis or risk of sepsis. Treatment with etanercept should not be initiated in patients with active infections (ie. hepatitis C, hepatitis B, active TBC)
* Is pregnant or breast-feeding
* Has significant concurrent medical diseases including, uncompensated congestive heart failure, myocardial infarction within 12 months, unstable angina pectoris, or history of human immunodeficiency virus (HIV) infection, immunodeficiency syndromes, or central nervous system (CNS) demyelinating events suggestive of multiple sclerosis
* Has a history of confirmed blood dyscrasias
* Received any live (attenuated) vaccines within 4 weeks of screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid Arthritis Patients, Psoriatic Arthritis Patients, Ankylosing Spondylitis Patients
Sampling Method: Non-Probability Sample
Enrollment: 880 (Actual)
Dates: Start 2006-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- Greece (6):
  - Pfizer Investigational Site, Thessaloniki, Asvestohori
  - Pfizer Investigational Site, Athens, Maroussi
  - Pfizer Investigational Site, Athens
  - Pfizer Investigational Site, Karditsa
  - Pfizer Investigational Site, Larissa
  - Pfizer Investigational Site, Thessaloniki

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A-101695&StudyName=Study%20Evaluating%20%20the%20Safety%20of%20Etanercept%20in%20Rheumatoid%20Arthritis%2C%20Ankylosing%20Spondylitis%20and%20Psoriatic%20Arthritis

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: Etanercept administered subcutaneously (s.c.) at a dose of 25 milligram (mg) twice weekly or 50 mg once weekly for 24 months.
Period: Overall Study
Arm/Group | Etanercept
Started | 880
Completed | 343
Not Completed | 537
Not completed — Not completed 24 month observation time | 334
Not completed — Lost to Follow-up | 101
Not completed — Withdrawal by Subject | 21
Not completed — Adverse Event | 81

BASELINE CHARACTERISTICS:
Arm/Group | Etanercept
Number analyzed (Participants) | 880
Age Continuous [Mean (Standard Deviation); unit: Years] — Mean age of the participants is based on N=795.
  Years | 52.0 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 562
  Male | 318

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Any untoward medical occurrence in a participant who received study drug was considered an AE, without regard to possibility of causal relationship. An AE resulting in any of the following outcomes, or deemed to be significant for any other reason, was considered to be a SAE: death; initial or prolonged inpatient hospitalization; a life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to Month 24
Population: Safety population included all participants who received at least one dose of etanercept.
Measure: Number; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 880
Participants
  AEs | 455
  SAEs | 36

2. Primary Outcome: Number of Participants Who Discontinued Treatment
Time Frame: Baseline up to Month 24
Population: Safety population included all participants who received at least one dose of etanercept.
Measure: Number; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 880
Participants | 203

3. Primary Outcome: Number of Participants by Reasons for Discontinuation of Treatment
Time Frame: Baseline up to Month 24
Population: Safety population included all participants who received at least one dose of etanercept.
Measure: Number; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 880
Participants
  Lost to follow-up | 101
  Withdrawal by participants | 21
  AEs | 60
  SAEs | 21

4. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ) at 24 Month
Description: HAQ is a measure of functional limitations. Participants were rated on 4 point scale with scores as 'normal' (no difficulty=0), 'adequate' (some difficulty= 1), 'limited' (much difficulty=2), and 'unable to do' (=3) based on degree of difficulty they experienced with 20 tasks grouped into 8 areas of dressing, rising, hygiene, reach, walking, eating, grip and activities. HAQ total scores were expressed as overall mean score ranging from 0 to 3: 0-0.25=normal functioning; 0.25-0.5=mild functional limitation; 0.5-1=moderate functional limitation; greater than 1=significant functional limitation.
Time Frame: Baseline, Month 24
Population: Data was not analyzed as the usage of the questionnaire was not considered to be part of usual clinical practice at the time of the study and thus was not to be used in the framework of a non-interventional trial.
Measure: Number; unit: Units on a Scale
Arm/Group | Etanercept
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline in Patient Global Assessment (PtGA) Visual Analog Scale (VAS) at 24 Month
Description: PtGA measured using a 100 mm VAS ranging from 0 = very good to 100 = very bad.
Time Frame: Baseline, Month 24
Population: Data was not analyzed as the usage of the scale was not considered to be part of usual clinical practice at the time of the study and thus was not to be used in the framework of a non-interventional trial.
Measure: Number; unit: Millimetre (mm)
Arm/Group | Etanercept
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in Physician Global Assessment (PGA) VAS at 24 Month
Description: PGA was measured on a 0 to 100 mm VAS, with 0 mm = no disease activity to 100 mm = worst disease activity possible.
Time Frame: Baseline, Month 24
Population: as for outcome 5
Measure: Number; unit: mm
Arm/Group | Etanercept
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 36/880
Other Adverse Events (participants affected / at risk) | 455/880
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept (N=880)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Uveitis (Eye disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Tooth abscess (Gastrointestinal disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Transaminases increased (Investigations) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 (3)
Suicide attempt (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Pyelonephritis (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Salpingitis (Reproductive system and breast disorders) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung neoplasm malignant (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia universalis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1)
Parathyroidectomy (Surgical and medical procedures) | 1 (1)
Thyroidectomy (Surgical and medical procedures) | 2 (2)
Lymphoedema (Vascular disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept (N=880)
Anaemia (Blood and lymphatic system disorders) | 21 (24)
Infectious mononucleosis (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 11 (14)
Leukopenia (Blood and lymphatic system disorders) | 8 (9)
Lymphocytosis (Blood and lymphatic system disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 5 (5)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytosis (Blood and lymphatic system disorders) | 3 (3)
Angina unstable (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Oedema peripheral (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Cushing's syndrome (Endocrine disorders) | 3 (3)
Conjunctivitis (Eye disorders) | 2 (2)
Dry eye (Eye disorders) | 3 (3)
Iridocyclitis (Eye disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 2 (2)
Aptyalism (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (5)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1)
Gastric infection (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 8 (8)
Gastroenteritis viral (Gastrointestinal disorders) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Asthenia (General disorders) | 3 (3)
Chest discomfort (General disorders) | 1 (1)
Chest pain (General disorders) | 3 (3)
Condition aggravated (General disorders) | 1 (1)
Discomfort (General disorders) | 1 (1)
Drug ineffective (General disorders) | 43 (43)
Fatigue (General disorders) | 2 (5)
Gait disturbance (General disorders) | 1 (1)
Injection site erythema (General disorders) | 13 (25)
Injection site irritation (General disorders) | 1 (1)
Injection site pain (General disorders) | 3 (9)
Injection site pruritus (General disorders) | 1 (1)
Injection site rash (General disorders) | 3 (3)
Injection site reaction (General disorders) | 7 (18)
Local reaction (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 3 (4)
Pyrexia (General disorders) | 2 (2)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 24 (25)
Hypertransaminasaemia (Lab Technical Error) (Hepatobiliary disorders) | 1 (1)
Peliosis hepatis (Hepatobiliary disorders) | 1 (1)
Drug eruption (Immune system disorders) | 1 (1)
Eyelid oedema (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2)
Urticaria (Immune system disorders) | 4 (8)
Febrile infection (Infections and infestations) | 4 (4)
Herpes ophthalmic (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Oral fungal infection (Infections and infestations) | 2 (2)
Oral herpes (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2)
Pilonidal cyst (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 27 (44)
Sinusitis (Infections and infestations) | 1 (2)
Soft tissue infection (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 6 (6)
Urinary tract infection (Infections and infestations) | 11 (14)
Vaginal infection (Infections and infestations) | 2 (2)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase decreased (Investigations) | 9 (9)
Alanine aminotransferase increased (Investigations) | 50 (56)
Anti-HBs antibody positive (Investigations) | 1 (1)
Aspartate aminotransferase decreased (Investigations) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 7 (7)
Basophil count decreased (Investigations) | 1 (1)
Basophil count increased (Investigations) | 1 (1)
Blood alkaline phosphatase decreased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 13 (18)
Blood calcium increased (Investigations) | 2 (2)
Blood calcium increased (Lab Technical Error) (Investigations) | 1 (1)
Blood cholesterol decreased (Investigations) | 14 (14)
Blood cholesterol increased (Investigations) | 88 (97)
Blood creatinine decreased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 9 (10)
Blood glucose decreased (Investigations) | 5 (5)
Blood glucose increased (Investigations) | 17 (17)
Blood phosphorus increased (Investigations) | 3 (3)
Blood phosphorus increased (Lab Technical Error) (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
Blood potassium increased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 4 (4)
Blood pressure systolic decreased (Investigations) | 1 (1)
Blood sodium increased (Investigations) | 2 (2)
Blood triglycerides decreased (Investigations) | 5 (5)
Blood triglycerides increased (Investigations) | 46 (50)
Blood urea decreased (Investigations) | 1 (1)
Blood urea increased (Investigations) | 17 (18)
Blood urine present (Investigations) | 2 (2)
C-reactive protein increased (Investigations) | 2 (2)
Differential white blood cell count abnormal (Investigations) | 35 (40)
Eosinophil count increased (Investigations) | 2 (3)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Haematocrit decreased (Investigations) | 4 (4)
Haematocrit normal (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 5 (5)
Hepatic enzyme increased (Investigations) | 2 (2)
High density lipoprotein decreased (Investigations) | 2 (2)
High density lipoprotein increased (Investigations) | 1 (1)
Low density lipoprotein decreased (Investigations) | 4 (4)
Low density lipoprotein increased (Investigations) | 15 (17)
Lymphocyte count decreased (Investigations) | 3 (3)
Lymphocyte count increased (Investigations) | 3 (3)
Monocyte count increased (Investigations) | 1 (1)
Neutrophil count increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 5 (5)
Platelet count increased (Investigations) | 3 (3)
Red blood cell count decreased (Investigations) | 1 (1)
Red blood cell sedimentation rate increased (Investigations) | 7 (11)
Transaminases decreased (Investigations) | 6 (6)
Transaminases increased (Investigations) | 9 (9)
Weight decreased (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 3 (3)
White blood cell count increased (Investigations) | 3 (3)
White blood cell count normal (Investigations) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 7 (7)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 11 (12)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3)
Hyperlipidaemia (Metabolism and nutrition disorders) | 18 (18)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4)
Iron deficiency anaemia (Metabolism and nutrition disorders) | 2 (2)
Oedema peripheral (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (25)
Arthritis (Musculoskeletal and connective tissue disorders) | 19 (21)
Arthropathy (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Demyelination plaque (Musculoskeletal and connective tissue disorders) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Finger deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3)
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 18 (28)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 6 (11)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 3 (3)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 9 (9)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 2 (2)
Synovial disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 10 (15)
Tendonitis (Musculoskeletal and connective tissue disorders) | 4 (5)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gallbladder polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3)
Head titubation (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 7 (7)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Hypoaesthesia facial (Nervous system disorders) | 1 (1)
Vertigo (Nervous system disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Emotional disorder (Psychiatric disorders) | 1 (1)
Fear of disease (Psychiatric disorders) | 1 (1)
Somnolence (Psychiatric disorders) | 1 (2)
Escherichia urinary tract infection (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 2 (2)
Breast mass (Reproductive system and breast disorders) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 1 (1)
Genital rash (Reproductive system and breast disorders) | 1 (1)
Libido disorder (Reproductive system and breast disorders) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (2)
Prostatitis (Reproductive system and breast disorders) | 5 (7)
Acute tonsillitis (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
H1N1 influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory tract infection viral (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tonsillitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (3)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 3 (4)
Erythema (Skin and subcutaneous tissue disorders) | 7 (11)
Nail psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Onychomycosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (10)
Psoriasis (Skin and subcutaneous tissue disorders) | 9 (16)
Rash (Skin and subcutaneous tissue disorders) | 10 (13)
Rash papular (Skin and subcutaneous tissue disorders) | 2 (2)
Rash pustular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Skin striae (Skin and subcutaneous tissue disorders) | 2 (2)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Tinea versicolour (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Contusion (Vascular disorders) | 3 (5)
Hypertension (Vascular disorders) | 7 (8)
Hypotension (Vascular disorders) | 1 (1)
Peripheral coldness (Vascular disorders) | 1 (1)
Venous insufficiency (Vascular disorders) | 1 (1)
(localized) arthritis (General disorders) | 4 (4)
acute sciatica and lumbago (General disorders) | 1 (1)
Breast tumor (General disorders) | 1 (1)
Decreased morning stiffness (General disorders) | 1 (2)
deformities of upper limbs bilaterally (General disorders) | 1 (1)
elbow Psoriasis (General disorders) | 1 (1)
hip arthritis (General disorders) | 1 (1)
hip pain and restriction of mobility (General disorders) | 1 (1)
Hypothermic lower limbs without pulse (General disorders) | 1 (1)
Improvement of spine mobility (General disorders) | 1 (1)
Increased inflammatory markers (General disorders) | 1 (1)
injury of gluteal muscle (General disorders) | 1 (1)
jaundice (biliary cirrhosis) (General disorders) | 1 (1)
joint pain, enthesitis (General disorders) | 1 (1)
localized nettle rash (General disorders) | 1 (1)
localized tender joints (General disorders) | 8 (12)
Lower limb deformities (General disorders) | 1 (1)
Measurement of the thoracic cage (General disorders) | 1 (1)
Mild conjunctivitis (General disorders) | 1 (1)
mild synovitis (General disorders) | 1 (1)
mobile, painful axillary lymph node (General disorders) | 1 (1)
Oligoarthritis (General disorders) | 1 (1)
Pain and restriction of mobility (General disorders) | 1 (1)
Paresthetic thigh pain (General disorders) | 1 (1)
pelvic fracture (fall) (General disorders) | 1 (1)
pelvic restriction of mobility (General disorders) | 1 (1)
Permanent disability in hand (General disorders) | 2 (2)
Plantar aponeurosis (General disorders) | 1 (1)
possible carpal tube syndrome (General disorders) | 1 (1)
relapsed rash psoriasiform (General disorders) | 1 (1)
Remission of scalp psoriasis (General disorders) | 1 (1)
restriction of hip mobility (General disorders) | 1 (1)
Restriction of movement of thoracic cage (General disorders) | 1 (1)
Restriction of shoulder mobility bilaterally (General disorders) | 1 (1)
Scalp pruritus (General disorders) | 1 (1)
sciatica and lumbago (General disorders) | 2 (2)
secondary osteoarthritis (General disorders) | 1 (1)
Shrinkage of tendon (General disorders) | 1 (1)
Swollen joints with restriction of mobility (General disorders) | 1 (1)
synovitis of limbs (General disorders) | 1 (1)
tender and swollen joints (General disorders) | 1 (2)
tender hip (General disorders) | 1 (2)
tender joints of lower limb (General disorders) | 1 (1)
tender spine (General disorders) | 2 (2)
Unstable gait (General disorders) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Wyeth has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.